CLINICAL TRIAL: NCT04181164
Title: Evaluation of Bone Architecture and Bone Strength in Adults With Hypophosphatasia (HPP)
Acronym: BABS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Nicola Hepp, Principal Investigator, MD, Hvidovre University Hospital
Other Study IDs: HvH-BABS-Study
Record Dates: First submitted 2019-11-18; First posted 2019-11-29 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Hypophosphatasia (HPP)
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HPP-Group: Adults with hypophosphatasia.
  Interventions: Other: Microindentation; Other: High resolution peripheral quantitative computed tomography (HRpQCT); Biological: Biochemical analysis of different bone markers.
- Control-Group: Healthy control subjects.
  Interventions: Other: Microindentation; Other: High resolution peripheral quantitative computed tomography (HRpQCT); Biological: Biochemical analysis of different bone markers.

INTERVENTIONS:
Other: Microindentation — Microindentation is a new technology directly measuring bone strength by a minimal invasive technique.
Other: High resolution peripheral quantitative computed tomography (HRpQCT) — HRpQCT scan can assess the cross-sectional geometry of the bone and is an appropriate investigation to evaluate bone quality.
Biological: Biochemical analysis of different bone markers. — Measurement of different bone markers by biochemical analysis of blood samples.

SUMMARY:
The study aims to evaluate the bone architecture and bone strength in adults with Hypophosphatasia (HPP).

ELIGIBILITY:
Inclusion criteria HPP-Group:

* Genetically verified HPP
* Age: ≥ 18 years
* Persistently low levels of alkaline phosphatase (ALP) ≤ 35 U/L (normal range 35-105 U/L)
* At least one of the following symptoms: a) dental manifestations; b) musculoskeletal pain; c) history of fracture(s)
* Submitted informed consent

Inclusion Criteria Control-Group:

* No ALP measurements ≤ 45 U/l and ≥ 50% of all ALP measurements, registered in the electronical clinical journal ≥ 55 U/l
* Normal parathyroid hormone (PTH) and Pyridoxal-5´-phosphate (PLP)
* Vitamin D3 ≥ 25 nmol/L
* Submitted informed consent

Exclusion criteria HPP-Group:

* Pregnancy
* Skin infection or severe skin affection in the measurement area of microindentation
* Known allergy to Lidocain
* Former or current medical treatment influencing bone metabolism (oral corticosteroid > 12 weeks, former or current anti-osteoporosis treatment at any time (regardless drug holiday), all kind of sex steroids (excluding oral contraception), anti-convulsants)
* Current malignant disorders

Exclusion Criteria Control-Group:

* Family history of a genetic metabolic bone disease (HPP, Osteogenesis imperfecta)
* Rickets in childhood
* Former or current Osteoporosis
* Former or current Osteomalacia
* Known diabetes
* Former or current medical treatment influencing bone metabolism (oral corticosteroid > 12 weeks, former or current anti-osteoporosis treatment at any time (regardless drug holiday), all kind of sex steroids (excluding oral contraception), anti- convulsants)
* Skin infection or severe skin affection in the measurement area of microindentation
* Chronic liver or gallbladder disease
* Current malignant disorders
* Former or current thyrotoxicosis (T4 over normal range ≥ 6 months)
* Cushing disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults, diagnosed with HPP (genetic verified) (n=15), matched 1:1 in case of gender, age (± 5 years), BMI (± 3 kg/m2), postmenopausal status (± 2 years) with healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Differences in Bone Mineral Strength Index (BMSi) between the two groups, assessed by microindentation (OsteoProbe®). | 1. October 2019 - 31.July 2020
  Differences in BMSi between the HPP- and Control-Group will be evaluated by microindentation (OsteoProbe®).
  Microindentation is a technology directly measuring bone strength by a minimal invasive technique. By applying a standardized pressure with a probe, which at the same time measures the indentation depth in the tibia bone, a measure of bone strength is obtained and calculated as Bone Mineral Strength Index (BMSi) [1].

SECONDARY OUTCOMES:
Correlation between BMSi and fracture prevalence in the HPP-Group and the Control-Group. | 1. October 2019 - 31.July 2020
  BMSi will be evaluated by microindentation (described above). In addition, information about the occurrence of fractures in the HPP- and Control-Group will be obtained by data from the Danish National Patient Register and a structured clinical interview.
Evaluation of differences in bone microarchitecture between the HPP- and Control-Group by high resolution peripheral quantitative computed tomography (HRpQCT). | 1. October 2019 - 31.July 2020
  To asses differences in bone architecture between the two groups, the non-dominant distal radius and non-dominant distal tibia will be examined by HRpQCT, which will provide data about total, trabecular and cortical BMD, trabecular thickness, cortical thickness, trabecular number, stiffness and finite element failure load of the radius and tibia.
Evaluation of differences in bone homeostasis between the two groups by biochemical analysis of different bone markers (P1NP, CTx, BALP, Trab-5, Sclerostin, Osteocalcin and FGF23) | 1. October 2019 - 31.July 2020
  Blood samples will be collected for biochemical analysis of different bone markers (P1NP, CTx, BALP, Trab-5, Sclerostin, Osteocalcin and FGF23).
  BALP = Bone specific alkaline phosphatase CTx = Carboxy-terminal collagen crosslinks FGF-23 = Fibroblast growth factor 23 P1NP = Procollagen type 1 amino-terminal propeptide Trab-5 = Tartrate-resistant acid phosphatase-5

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrera S, Diez-Perez A. Clinical experience with microindentation in vivo in humans. Bone. 2017 Feb;95:175-182. doi: 10.1016/j.bone.2016.11.003. Epub 2016 Nov 11. PMID 27840302